CLINICAL TRIAL: NCT03470090
Title: Assessment Effects of Neuromuscular Exercises Training on Physical Activity, Functionality and Balance in Knee Osteoarthritis
Brief Title: The Effects of Neuromuscular Exercises Training on Physical Activity, Functionality and Balance in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Asistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/72
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Exercise; Osteoarthritis
Keywords: Physical activity; Function; Balance; Neuromuscular exercises; Osteoarthritis
MeSH Terms: conditions — Motor Activity; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Who Masked: Participant
Masking Description: Participants didn't know taking which exercise treatment methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Exercises Group (Experimental): This group of patients received patient with knee osteoarthritis. It will be applied classical physiotherapy and neuromuscular exercises training
  Interventions: Behavioral: Neuromuscular Exercises
- Conventional Group (Active Comparator): This group of patients received patient with knee osteoarthritis. It will be applied classical physiotherapy and conventional exercises.
  Interventions: Behavioral: Conventional Group

INTERVENTIONS:
Behavioral: Neuromuscular Exercises — In the experimental group, the subjects who were taken into the study were taken to the neuromuscular exercise (NME) program after the pre-treatment evaluations. The subjects in this group were given classical physiotherapy and NME performed 6 days a week, 1 set of 10 times physiotherapist control. NME was including warming, neuromuscular exercises (balance, muscle strengthening, proprioception, sensorimotor system training, joint stabilization and postural control exercises) and cooling periods.
  Arms: Neuromuscular Exercises Group
Behavioral: Conventional Group — In the control group, the subjects who were taken into the study were taken to the classical physiotherapy (hotpack (HP), ultrasound (US), transcutaneous electrical stimulation (TENS)) and conventional exercises program after the pre-treatment evaluations.
  Arms: Conventional Group

SUMMARY:
This study was planned to evaluate the effect of neuromuscular exercise program on physical activity, functionality and balance in patients with knee osteoarthritis aged 35-65 years.

DETAILED DESCRIPTION:
The degeneration that occurs in the osteoarthritis of the knee joint leads to the loss of proprioception, resulting in the misalignment of the mechanoreceptors in that region, the joint stabilization is impaired, the muscles do not fulfill the protective role and the joint neuromuscular is inadequate for control. Neuromuscular control is the subcortical activity of effector structures against stimulation with mechanoreceptor, visual, and vestibular affinities. Proprioception, kinesthesia, sensation of joint position, visual and vestibular information constitute sensory data; functional motor patterns, dynamic joint stability and reactive neuromuscular control motor efferent response definitions. Disturbance of neuromuscular control of the muscles also affects walking and balance with abnormal weight transfer. There are many ways to treat knee osteoarthritis such as patient education, weight control, different physical therapy modalities (hot, cold, electrotherapy, deep heat), exercise, pharmacological treatments (topical, systemic, intraarticular). There is no radical treatment of osteoarthritis to restore structural changes; but with the treatment applied, findings such as pain and loss of function of the individual can be reduced and the patients become more independent in daily life activities. Surgical treatment is the last resort in osteoarthritis. In osteoarthritis( OA), there is no pharmacological method to treat the deformed joint structure that will change the course of the disease. This situation significantly increases the importance of rehabilitation in the treatment of osteoarthritis. The aim of neuromuscular rehabilitation that reestablish and regulated features such as dynamic joint stability, reactive neuromuscular control, functional motor patterns. Rehabilitation programs created for this purpose include balance exercises, strengthening exercises, postural control, functional exercises, postural orientation, flexibility, agility, plyometric exercises, spore-specific exercises. neuromuscular exercise program includes 7 parameters including functional mobility, functional stability, sensorimotor system training, proprioceptive neuromuscular facilitation training techniques, plyometric exercises, reactive neuromuscular system training, technical training. Main purpose of this study is that the effect of neuromuscular exercise program on physical activity, functionality and balance in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis,
* individuals without a physical disability,
* person in an age range 35- 65 years,
* Having no any knee surgeon,
* Mentally that is sufficient to make assessments,
* Who want to be involved voluntary work,
* Ability to adjust the training program
* Individuals who received informed consent

Exclusion Criteria:

* Individuals who do not allow mental evaluation
* Individuals who do not want to be involved in voluntary work.
* Clinical study refused to participate in.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-16 (Actual)

PRIMARY OUTCOMES:
Change from Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) of patients with knee osteoarthritis at 6 weeks. | 6 weeks
  The scale used to measure knee function (0-100 total score). High scores indicate poor function status and low scores indicate good function status. The scale contains 24 questions, three subgroups of pain, stiffness and physical function.
  There are 5 alternative answers to the questions: 0 = no, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe The rating (total of all answers / 96) was calculated as * 100.

SECONDARY OUTCOMES:
Changed from Visual Analog Scale (VAS) of patients with knee osteoarthritis at 6 weeks. | 6 weeks
  It used to measure level of pain (0-100 mm). On a horizontal line of 100 millimeters (mm), the initial 0 (no pain) and end (pain at unbearable grade) were marked. It was requested to place a mark on this horizontal line according to the degree of pain they felt in the cases. The point marked on the line was then recorded as a VAS value in mm, measured by a ruler.
Change from International Physical Activity Questionnaire (IPAQ) Short Form of patients with knee osteoarthritis at 6 weeks. | 6 weeks
  It used to measure level of physical activity. IPAQ short form; 7 questions that provide information about time spent on walking, moderate to severe activities, and time spent sitting. The energy required for the activities was calculated by the MET-minute score. Standard MET values for these activities are: Walk = 3,3 MET; Moderate Severe Physical Activity = 4,0 MET; Severe Physical Activity = 8.0 MET; Seating = 1,5 MET.
Change from Y Balance Test of patients with knee osteoarthritis at 6 weeks. | 6 weeks
  It used to measure static balance.Anterior (A), Posteromedial (PM) and posterolateral (PL) measurements were performed. It was glued to three graves at 120 degrees. The patient was asked to put one foot on the intersection of these three bombers and to lie in directions A, PM, and PL with the other foot. During the test, the patient was asked to point to the maximum point he could reach without touching his foot and to bring it to the stable foot without losing balance. The distance is measured in centimeters.
Change from 2000 International Knee Documentation Committee (IKDC) of patients with knee osteoarthritis at 6 weeks. | 6 weeks
  It used to measure functionality.
  The questionnaire consists of 10 questions in total. 0 is the worst level of activity when measuring activity level; 4 is answered for the maximum level of activity. Similarly, when evaluating frequency, 0 is the most severe, 10 is not. 0-100 total score.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Talu, PhD, Principal Investigator — Inonu University
Locations (1):
- Malatya Gozde Hospital, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No